CLINICAL TRIAL: NCT01737476
Title: Trial to Evaluate the Efficacy of the HLPFC Coil Deep Transcranial Magnetic Stimulation System in Treating Attention Deficit and Hyperactivity Disorder (ADHD) in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sor010912ctil
Record Dates: First submitted 2012-09-20; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Attention Deficit Disorder Patients
Keywords: age 18-65

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- control (Sham Comparator): control-sham
  Interventions: Procedure: Transcranial Magnetic Stimulation. PFC
- Deep TMS PFC Lt (Active Comparator): Deep TMS PFC left
  Interventions: Procedure: Transcranial Magnetic Stimulation. PFC
- DEEP TMS PFC Rt (Active Comparator): DEEP TMS PFC Rt
  Interventions: Procedure: Transcranial Magnetic Stimulation. PFC
- Superficial TMS PFC Lt (Active Comparator): Superficial TMS PFC Lt
  Interventions: Procedure: Transcranial Magnetic Stimulation. PFC
- superficial TMS PFC Rt (Active Comparator): superficial TMS PFC Rt
  Interventions: Procedure: Transcranial Magnetic Stimulation. PFC

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation. PFC
  Other Names: Stimulator: Magstim rapid2. The Magstim Company Limited, Spring gardens, Whitland, Carmarthenshire, SA34 OHR, UK.; Coil: HLPFC. Brainsway Ltd. 19 hartum St. Bynet Building, Har Hatzofim, Jerusalem, Israel.

SUMMARY:
The aim of the study is to investigate the efficacy of trans-cranial magnetic stimulation in treating attention deficit disorder in adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* ADD/ADHD

Exclusion Criteria:

* any DSM-IV psychiatric disorder except ADD/ADHD
* use of psychoactive medications
* Epilepsy
* brain injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ben-Gurion University, Beersheba, Israel

REFERENCES:
- [Derived] Hadas I, Hadar A, Lazarovits A, Daskalakis ZJ, Zangen A. Right prefrontal activation predicts ADHD and its severity: A TMS-EEG study in young adults. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Dec 20;111:110340. doi: 10.1016/j.pnpbp.2021.110340. Epub 2021 May 3. PMID 33957168